CLINICAL TRIAL: NCT02683590
Title: STernectOmy Repair Efficiency of a Ceramic Implant
Acronym: STOIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: I15032
Record Dates: First submitted 2016-02-02; First posted 2016-02-17 (Estimated); Last update posted 2019-08-12 (Actual); Status verified 2017-01

CONDITIONS: Bones, Tumors
Keywords: Sternectomie; Ceramic Implant; Bones Tumors
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sternum by a ceramic implant (Experimental): The replacement of the sternum by a ceramic implant
  Interventions: Device: Ceramic Implant

INTERVENTIONS:
Device: Ceramic Implant — The replacement of the sternum by a ceramic implant

SUMMARY:
For the replacement of the sternum, there is no consensus regarding the most appropriate and most effective physiologically material. The use of ceramic implant offers significant operational time saving and biocompatibility coupled with the strength of the material allow us to realize a more natural operation, limiting the risk of infection and rejection.

Main objective: to evaluate the efficiency of the replacement of the sternum by a ceramic implant on the respiratory capacity at 3 months post surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient major
* Having a replacement indicating the sternum (or a part of the sternum)
* With an expected life of over one year, estimated by the principal investigator
* Written consent of the patient

Exclusion Criteria:

* People under safeguard justice,
* Patient under guardianship,
* Patient pregnant or breastfeeding,
* Topic attending another search including a period of exclusion still going to run-in
* Contraindication to general anesthesia
* Of alumina allergy antecedent
* Recent infectious disease unsupported
* BMI> 40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-03; Primary Completion 2019-05 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
vital capacity | 1 day
  Slow Vital Capacity (liters), forced vital capacity (liters)

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Limoges Hospital, Limoges
  - Saint George clinic, Nice
  - Reims university hospital, Reims

IPD SHARING:
Plan to Share IPD: No